CLINICAL TRIAL: NCT05229224
Title: Evaluation of the Efficacy of the Osteo-Fluidic-sensitive (OFS) Versus Placebo Method in the Management of Frequent Episodic Tension-type Headache. Pilot Study.
Brief Title: Pilot Study of the Osteo-Fluidic-Sensitive (OFS) in Tension-type Headache.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CephalOFS
Record Dates: First submitted 2022-01-26; First posted 2022-02-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-01

CONDITIONS: Tension-Type Headache Episodic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteo-Fluidic-Sensitive method (Experimental)
  Interventions: Other: Osteo fluidic Sensitive méthod
- Placebo method (Placebo Comparator)
  Interventions: Other: Placebo method

INTERVENTIONS:
Other: Osteo fluidic Sensitive méthod — Manual therapy, without manipulative treatment, based on rebalancing of the body with manual pressures on specific body areas.
  Arms: Osteo-Fluidic-Sensitive method
Other: Placebo method — Soft Manual pressures at specific points that are defined as non-effective and non-deleterious for patients.
  Arms: Placebo method

SUMMARY:
The hypothesis of the study is the Osteo-fluidic-Senstive is effective for lowering headache pains (Reduction of the number of days of headaches per month) for patients having frequent episodic tension-type headache. The OFS method will improve quality of life and will reduce the consumption of crisis treatments.

Compare the efficacy of the Osteo-Fluidic-Sensitive method versus a placebo method on patients with tension type headache for the reduction of the number of days of headaches per month after 3 months of treatment at Centre Hospitalier Universitaire de Poitiers.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 75 years' old
* Person having highly frequent episodic tension type headache (between 2 and 14 days of headaches per month) associated or not to headache with characteristic of a migraine per International Classification of Headache Disorders 3rd edition criteria
* Person who completed his headache agenda the month before the study.
* Patient who understands and accepts the effects of the study
* Signed consent
* Person with health insurance coverage

Exclusion Criteria:

* Person having secondary or primary headaches (chronic tension type headache, migraines only, Cluster headaches, Neuralgias ...)
* Person on treatment of venlafaxine, gabapentine, duloxetine, clomipramine et toxine botulique.
* Concomitant participation to another clinical research
* Pregnant or lactating women, women of child-bearing age who do not have effective contraception.
* People with reinforced protection (juvenile), people deprived of liberty per justice or administrative decision, people living in a sanitary and social establishment, adults under legal protection and people in critical medical conditions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-05-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
numbers of days with headaches | one month
  The main criteria for the study will be the difference of the number of days with headaches evaluated based on a calendar of headaches between the month prior to the beginning of the treatment and the month following the last session (1st month).

CONTACTS AND LOCATIONS:
Overall Officials: Helene KERSUZAN, Principal Investigator — CHU de Poitiers FRANCE
Locations (1):
- CHU Poitiers, Poitiers, France